CLINICAL TRIAL: NCT05418595
Title: Ultrasonographic Evaluation of Ovarian Stroma in PCOS Women
Brief Title: Ultrasonographic Evaluation of Ovarian Stromal Vascularity in Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Usak State Hospital (Other)
Responsible Party: Principal Investigator, Irem Senyuva, Usak Training and Research hospital, Usak State Hospital
Other Study IDs: 575704
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group-1: PCOS patients intraovarian stromal conventional and SMI doppler findings

INTERVENTIONS:
Other:

SUMMARY:
The most common endocrine condition in reproductive women is polycystic ovary syndrome. It has a prevalence of 5-10%. According to the Rotterdam criteria, oligo/anovulation, clinic or biochemical hyperandrogenism, PCOS morphology in ultrasonography, and the presence of these two criteria are required for diagnosis.

The echogenicity of the ovarian stroma, vascularity, ovarian size, cystic pattern density, and subcortical organization of cysts are all significant considerations in ultrasonographic evaluation.

DETAILED DESCRIPTION:
Retrospective archive study.

In the years 2018-2019, the ultrasonographic archives of PCOS women will be analyzed retrospectively in the Radiology department of Usak Education and Research Hospital. Ultrasonographic (Two-dimensional ultrasonography , conventional and other doppler) measurements of ovaries will be assessed in ultrasonographic data. Patient's data ( Menstrual cycle, androgenic findings, age, BMI etc..) will be obtained on the hospital records, PCOS patient's phenotype will be evaluated according to National Institutes Health (NIH) recommendations.

The ovarian ultrasonographic findings of PCOS women will be compared.

This study approved by Usak University Medical Faculty Ethical Committee April,06,2022.

The Ethical Committee decision number is 57-57-04.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive period According to Rotterdam criteria PCOS women.

Exclusion Criteria:

Women have not PCOS criteria, Non-reproductive period Pregnancy Postpartum Ovarian mass Underwent ovarian surgery.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive period, PCOS women
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
The superiority of Superb microvascular imaging doppler technique over the conventional doppler techniques | 1 month
  The Toshiba Aplio 500 ultrasonography tool (Toshiba, Aplio 500, Tokyo, Japan) was used in the Radiology Policlinic Ultrasonography Unit to perform ultrasonography using a 1-6 MHz convex probe. After scanning the lesion with TAUSG, 5-12 second-long video pictures were recorded. The ovarian stromal vascularity was defined according to the International Ovarian Tumor Analysis (IOTA) group criteria. Four categories of endometrial blood flow were identified: No coloration in grade 1, one or more punctate colorations in grade 2, one linear coloring or several (>5) punctate colorations in grade 3, and multiple linear colorations in grade 4 of the ovary. [14]. The vascularization rating was done independently using CDI, PDI, cSMI, and mSMI techniques. In all patients, the ovarian morphologic features were recorded for the both ovaries. Three radiologists analyzed the captured video pictures and assigned a consensus rating.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Şenyuva, MD, Principal Investigator — USAK TRAINING AND RESEARCH HOSPITAL, DEPARTMENT OF OBSTETRICS AND GYNECOLOGY,TURKEY
Locations (1):
- İrem Şenyuva, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozdemir O, Sari ME, Kalkan D, Koc EM, Ozdemir S, Atalay CR. Comprasion of ovarian stromal blood flow measured by color Doppler ultrasonography in polycystic ovary syndrome patients and healthy women with ultrasonographic evidence of polycystic. Gynecol Endocrinol. 2015 Apr;31(4):322-6. doi: 10.3109/09513590.2014.995617. Epub 2015 Jan 5. PMID 25558942
- [Background] Makled AK, El Sherbiny M, Elkabarity R. Assessment of ovarian stromal blood flow after metformin treatment in women with polycystic ovary syndrome. Arch Gynecol Obstet. 2014 Apr;289(4):883-91. doi: 10.1007/s00404-013-3057-8. Epub 2013 Nov 7. PMID 24196302